CLINICAL TRIAL: NCT00427544
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PRA-027 Administered Orally to Healthy Women of Nonchildbearing Potential
Brief Title: Study of the Safety, Tolerability, and PK of PRA-027 Administered to Women of Nonchildbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3208A1-1000
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Fibroid
Keywords: Uterine leiomyomata (Fibroids)
MeSH Terms: conditions — Leiomyoma; Myofibroma

INTERVENTIONS:
Drug: PRA-027

SUMMARY:
The primary purpose of this study is to asess the safety and tolerability of ascending single oral doses of PRA-027 in healthy women of nonchildbearing potential. The secondary purpose is to provide the initial pharmacokinetic (PK) and pharmacodynamic (PD) profile of PRA-027 in healthy women of nonchildbearing potential, and to evaluate the effect of a high-fat meal on the PK and PD of PRA-027 administered to healthy women of nonchildbearing potential.

ELIGIBILITY:
INCLUSION CRITERIA

* Women of nonchildbearing potential (WONCBP) aged 18 to 60 years. Must have a negative pregnancy test result within 48 hours before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or ultrasound scan.
* Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight ³50 kg. BMI is calculated by taking the subject's weight, in kilograms, divided by the square of the subject's height, in meters, at screening: BMI=weight (kg)/[height (m)]2
* Healthy as determined by the investigator on the basis of screening evaluations.

EXCLUSION CRITERIA

* Any significant cardiovascular, hepatic, renal, respiratory, gynecologic, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
* A history of drug abuse within 1 year before study day 1, a history of alcoholism within 1 year before study day 1 or consumption of more than 2 standard units of alcohol per day (a standard unit equals 12 ounces of beer, 1½ ounces of 80-proof alcohol, or 6 ounces of wine). Any positive findings during the urine drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, and opiates.
* Use of any investigational or prescription drug within 30 days before test article administration. Consumption of any caffeine-containing products (eg, coffee, tea, chocolate, or soda) or alcoholic beverages within 48 hours before study day 1. Consumption of grapefruit or grapefruit-containing products within 72 hours before study day 1. Use of any over-the-counter drugs, including herbal supplements (except for the occasional use of acetaminophen and vitamins ≤100% of the recommended daily allowance) within 14 days before study day 1.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-02; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to asess the safety and tolerability of ascending single oral doses of PRA-027 in healthy women of nonchildbearing potential.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Miami, Florida, United States